CLINICAL TRIAL: NCT01169051
Title: A Retrospective Analysis of Statin Use and Outcome After Thoracic Cancer Surgery
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 100698
Record Dates: First submitted 2010-07-14; First posted 2010-07-23 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Esophagectomy; Pulmonary Wedge Resection; Pulmonary Lobectomy; Pulmonary Pneumonectomy
Keywords: Esophagectomy; Pulmonary wedge resection; Pulmonary lobectomy; Pulmonary pneumonectomy; Thoracic Surgery; Lung Cancer; Esophageal Cancer
MeSH Terms: conditions — Lung Neoplasms; Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Thoracic sugery statins
- Thoracic surgery non-statins

SUMMARY:
There is data to support an association between impaired preoperative endothelial function and adverse postoperative outcome. This study will investigate the potential association between perioperative statin use and improved perioperative and long-term cancer outcome amongst thoracic surgery patients undergoing lung or esophageal resection.

DETAILED DESCRIPTION:
Statins are well established for the use of primary and secondary prevention of cardiovascular disease. Moreover, there is increasing evidence that statins have numerous effects separate from their lipid lowering properties-pleiotropic effects. These pleiotropic effects, including a reduction in the inflammatory response and improved endothelial function, may improve perioperative outcomes via modulation of the surgical stress response. Improved perioperative outcomes have been demonstrated in patients undergoing vascular, cardiac and non-cardiovascular surgery. Specific to the thoracic surgery population, statin use has been reported to reduce the incidence of atrial fibrillation.

Statins, via inhibition of the rate limiting step of the mevalonate pathway, have also sparked interest in their potential anticancer effects as well as in cancer prevention. There is some evidence for anticancer effects of statins in patients with esophageal and lung cancer. Additionally, other agents with known anti-inflammatory effects also point to the potential for improved outcome in cancer patients. In this regard, aspirin use is reported to associate with prolonged survival in breast cancer patients, while perioperative use of anti-inflammatory agents (COX-II inhibitor use and lung cancer; aprotinin use and mesothelioma; aprotinin use and esophageal cancer) is associated with improved postoperative survival. Moreover, the use of regional analgesia is commonly employed in the thoracic surgery population and has been associated with attenuation of metastasis and improvement in recurrence rates for some types of cancers.

In a prospective pilot study of patients undergoing elective thoracic surgery, a collaborative member of our group recently found that patients suffering postoperative complications had poorer endothelial function, as measured by flow mediated dilation. Those patients with poorer endothelial function had greater wound healing complications (6% vs. 0%, p=0.01), longer ICU length of stay (4 vs. 0.9 days, p=0.02), and longer hospital length of stay (14 vs. 6.9 days, p=0.01). Although this pilot study was underpowered to demonstrate a significant correlation between Brachial Artery Reactivity Testing (BART) derived endothelial function and "all" postoperative complications, it provides hypothesis generating data and supports the hypothesis that statins, as modulators of endothelial function, may have a role in improving postoperative outcome.

ELIGIBILITY:
Inclusion Criteria:

This study is a retrospective chart review of adult thoracic surgery patients who underwent:

* Esophagectomy
* Pulmonary wedge resection
* Pulmonary lobectomy
* Pulmonary pneumonectomy

Data collected will be from January 1, 2007 forward

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is a retrospective chart review of adult thoracic surgery patients who underwent:
  * Esophagectomy
  * Pulmonary wedge resection
  * Pulmonary lobectomy
  * Pulmonary pneumonectomy
  Data collected will be from January 1, 2007 forward.
Sampling Method: Non-Probability Sample
Enrollment: 569 (Actual)
Dates: Start 2010-07; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Effect of perioperative statin use on in-hospital morbidity after thoracic cancer surgery

SECONDARY OUTCOMES:
Effect of perioperative statin use on the development of Major Adverse Pulmonary Events (MAPE) | 30 days after initial surgery
  Includes acute lung injury, acute respiratory distress syndrome, pulmonary embolus, respiratory failure requiring mechanical ventilation and pneumonia
Effect of perioperative statin use and the development of Major Adverse Cardiac Events (MACE) | 30 days after initial surgery
  Includes atrial fibrillation, other arrhythmia, myocardial infarction and congestive heart failure.
Effect of perioperative statin on mortality associated with cancer recurrence following thoracic cancer surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Justin Sandall, D.O., Principal Investigator — Vanderbilt University; Mias Pretorius, M.D., Study Director — Vanderbilt University